CLINICAL TRIAL: NCT05901584
Title: A Single-arm Multicenter Phase II Clinical Trial of Cadunilumab (Anti-PD-1/CTLA-4) in Combination With or Without Chemotherapy in Second-line Treatment for Patients With Extensive Stage Small Cell Lung Cancer
Brief Title: Cadonilimab (AK104) With or Without CT as 2rd Line Treatment for ES-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Zunyi Medical University (Other)
Collaborators: Guizhou Provincial People's Hospital (Other); The First People's Hospital of Zunyi (Other); Guizhou Tongren People's Hospital (Unknown); The People"s Hospital of Xingyi (Unknown); The Second Affiliated Hospital of Guizhou Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SAHZunyiMU
Record Dates: First submitted 2023-06-04; First posted 2023-06-13 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Immunotherapy; Second-line Treatment
Keywords: Cardunilizumab; Small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (AK104) combined with chemotherapy (Experimental): Cadonilimab(10mg/kg, administered on the first day of each cycle, Q3W, until there is no clinical benefit)+platinum-based chemotherapy or Cadonilimab(10mg/kg, administered on the first day of each cycle, Q3W, until there is no clinical benefit), Q3W, 4cycles), every 3 weeks (21 days) is a treatment cycle
  Interventions: Drug: Cadonilimab

INTERVENTIONS:
Drug: Cadonilimab — Cadonilimab (10mg/kg, administered on the first day of each cycle, Q3W, until there is no clinical benefit)+platinum-based chemotherapy or Cadonilimab (10mg/kg, administered on the first day of each cycle, Q3W, until there is no clinical benefit), Q3W, 4cycles), every 3 weeks (21 days) is a treatment cycle.
  Other Names: AK104

SUMMARY:
This study is a phase II clinical study of Cadonilimab (AK104) combined with or without chemotherapy in the treatment of PD-1 inhibitor-resistant extensive stage small cell lung cancer

DETAILED DESCRIPTION:
This study is conducted by enrolling subjects with ES-SCLC who have previously failed first-line systemic therapy (platinum-containing chemotherapy in combination with or without atezolizumab and dulvalizumab), and all enrolled subjects will receive cadunilumab alone or in combination with chemotherapy and continue treatment in 3-week dosing cycles until toxicity is intolerable, there is no longer clinical benefit in the judgment of the investigator (in the investigator's judgment based on RECISTv1.1 imaging assessment and clinical status, etc.), completion of 24 months of treatment, or other criteria for termination of treatment in the protocol are met, whichever occurs first. Patients were observed for efficacy and side effects. Primary outcome: progression-free survival (PFS) based on RECIST v1.1 assessment. Secondary outcomes included: incidence and severity of adverse events; objective remission rate (ORR), disease control rate (DCR), duration of remission (DoR), time to remission (TTR), and overall survival (OS). Finally, mRNA expression profiles in tumor tissue samples were determined by gene sequencing to analyze the correlation between molecular subtypes of small cell lung cancer, immune-related gene characteristics and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in this study by signing an informed consent form.
2. Pathologically confirmed diagnosis of small cell lung cancer, with imaging confirmation of extensive stage with measurable lesions.
3. Patients who have been treated with at least one line of systemic platinum-containing chemotherapy regimen (with or without immunotherapy).

4.18 - 75 years of age; ECOG PS score: 0 to 1; expected survival greater than 3 months.

5.Major organ function within 7 days prior to treatment, meeting the following criteria:

* Blood test criteria (in 14-day untransfused state):

  1. Hemoglobin (HB) ≥ 90g/L.
  2. Absolute central granulocyte value (ANC) ≥ 1.5×109/L.
  3. Platelets (PLT) ≥75×109/L.

     ②Biochemistry needs to meet the following criteria:

  <!-- -->

  1. total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN).
  2. alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5 × ULN, if accompanied by liver metastases, then ALT and AST ≤ 5 × ULN
  3. serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance ≥ (CCr) 60 ml/min. ③Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ low limit of normal (50%).

     6.Female participants of reproductive age must use contraception methods such as IUD, pill, or condom during the study period and for 6 months after. Male participants must also agree to use contraception during the study period and for 6 months after. Additionally, female participants must have a negative serum or urine pregnancy test within 7 days prior to study entry and should not be breastfeeding.

     Exclusion Criteria:
     1. Patients with previous use of cardunilizumab.
     2. non-small cell lung cancer (including lung cancer with a mixture of small cell and non-small cell carcinoma).
     3. Patients with other types of cancer that occurred within the past 5 years or are currently present, with the exception of treated cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors that have not invaded the basement membrane (Ta, Tis, and T1).
     4. Systemic antitumor therapy, including cytotoxic therapy, signal transduction inhibitors, immunotherapy, within 4 weeks prior to enrollment or planned during the current study dosing period (or have used mitomycin C within 6 weeks prior to treatment with the trial drug). Have had extended field radiotherapy (EF-RT) within 4 weeks prior to subgroup or have had field-limited radiotherapy to the tumor lesion to be evaluated within 2 weeks prior to subgroup.
     5. Unremitted toxic reactions due to any prior treatment above CTCAE grade 1, excluding alopecia and neurotoxicity ≤ grade 2 due to oxaliplatin.
     6. Individuals with various factors such as difficulty swallowing, chronic diarrhea, and intestinal obstruction may experience challenges with oral drug administration.
     7. with pleural effusion or ascites causing respiratory syndrome (≥ CTCAE grade 2 dyspnea).
     8. Patients with brain metastases with symptoms or symptoms controlled for less than 2 months.
     9. Patients with any severe and/or uncontrolled disease, including:

  <!-- -->

  1. Patients with poorly controlled blood pressure (systolic blood pressure ≥ 150 mmHg and diastolic blood pressure ≥ 100 mmHg).
  2. Patients with myocardial ischemia of grade I or higher, myocardial infarction, arrhythmias (including QTc ≥ 480 ms), and congestive heart failure of grade 2 or higher (categorized according to the New York Heart Association (NYHA) classification) are included.
  3. Active or uncontrolled serious infection (≥ CTC AE grade 2 infection).
  4. Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis requiring antiviral therapy.
  5. Renal failure requiring hemodialysis or peritoneal dialysis.
  6. This refers to a medical history of immunodeficiency, which can be acquired through HIV or other diseases, or congenital in nature. It also includes a history of organ transplantation.
  7. poorly controlled diabetes (fasting blood glucose (FBG) >10 mmol/L).
  8. urine routine suggesting urine protein ≥++ and confirmed 24-hour urine protein quantification >1.0 g.
  9. Patients with seizures and requiring treatment. 10. Participants who have undergone major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of the study will be excluded.

     11.Patients whose imaging shows that the tumor has invaded the critical vascular perimeter or who, in the judgment of the investigator, are at high risk of fatal hemorrhage due to tumor invasion of a critical vessel during the follow-up study.

     12.Patients with any physical signs or history of bleeding, regardless of severity; patients with any bleeding or hemorrhagic event ≥ CTCAE grade 3, unhealed wounds, ulcers or fractures within 4 weeks prior to subgroup.

     13.Individuals who have experienced an arterial or venous thrombotic event within the past 6 months, including cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolisms, should take caution.

     14.Individuals with a history of psychotropic substance abuse or psychiatric disorders who are unable to abstain.

     15.having participated in clinical trials of other antineoplastic drugs within four weeks.

     16.Patients with concomitant diseases that are deemed to pose a significant risk to their safety or may hinder their ability to complete the study, as determined by the investigator, will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival，PFS | Time Frame: The last subject completes at least 24 weeks of follow-up (or disease progression)
  The time from the beginning of the patient's treatment to the disease progression or death for any reason.Based on RECIST v i I Assessed PFS

SECONDARY OUTCOMES:
Overall Survival,OS | 3 years
  The time from the patient receiving treatment to the death of the patient for any reason,OS evaluated according to RECIST vi. I
Objective Response Rate，ORR | The last subject completes at least 24 weeks of follow-up (or disease progression)
  The proportion of patients whose tumor volume is reduced to 30% and can be maintained for more than 4 weeks,Based on RECIST v i I Assessed ORR
Disease control rate,DCR | The last subject completes at least 24 weeks of follow-up (or disease progression
  Includes complete remission, partial remission, and stable disease maintained for more than 4 weeks as a percentage of patients with evaluable outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Hu Ma, Ph.D, Principal Investigator — The Second Affiliated Hospital of Zunyi Medical University
Locations (1):
- The Second Affiliated Hospital of Zunyi Medical University, Guizhou, ZunYi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pang X, Huang Z, Zhong T, Zhang P, Wang ZM, Xia M, Li B. Cadonilimab, a tetravalent PD-1/CTLA-4 bispecific antibody with trans-binding and enhanced target binding avidity. MAbs. 2023 Jan-Dec;15(1):2180794. doi: 10.1080/19420862.2023.2180794. PMID 36872527
- [Derived] Chen C, Chen M, Bai Y, Li Y, Peng J, Yao B, Feng J, Zhou JG, Ma H. A Single-Arm Multi-Center Phase II Clinical Trial of Cadonilimab (anti-PD-1/CTLA-4) in Combination with or without Conventional Second-Line Treatment for Patients with Extensive Stage Small Cell Lung Cancer. Technol Cancer Res Treat. 2024 Jan-Dec;23:15330338241249690. doi: 10.1177/15330338241249690. PMID 38706247